CLINICAL TRIAL: NCT02305498
Title: Yoga Practice for Breast or Ovarian Cancer Patients: A Pilot Study
Brief Title: Yoga Practice for Breast or Ovarian Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-059
Record Dates: First submitted 2014-11-25; First posted 2014-12-02 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: Yoga; 14-059
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms

ARMS (2):
- Vigorous yoga practice (Experimental): Supervised vigorous yoga practice, 60 minutes/session, 3 sessions/wk for 12 weeks, followed by 12 weeks of home practice.
  Interventions: Other: Vigorous yoga practice
- Restorative (gentle) yoga practice (Active Comparator): Supervised restorative (gentle) yoga practice, 60 minutes/session, 3 sessions/wk for 12 weeks, followed by 12 weeks of home practice.
  Interventions: Other: Restorative (gentle) yoga practice

INTERVENTIONS:
Other: Vigorous yoga practice
  Arms: Vigorous yoga practice
Other: Restorative (gentle) yoga practice
  Arms: Restorative (gentle) yoga practice

SUMMARY:
Previous research suggests that regular physical activity may make cancer survivors do better in the long run. Laboratory studies suggest that stress may be bad for cancer patients as well. The investigators are interested in whether yoga, a practice that combines physical activity and stress reduction, is beneficial to cancer survivors. To answer that question, the investigators will need to do a large scale clinical trial.

Before the investigators can do that large study, they need to know whether people are willing to participate in this kind of study, whether they can do the yoga practice regularly and for how long, what kind of changes they may experience in how they can handle their daily activities, emotion, sleep, memory and problem solving ability, and what are the changes that can happen in their body after doing the yoga practice. Answering these questions is what this study is about.

ELIGIBILITY:
Inclusion Criteria:

* Woman age 18 or older
* History of stage 0-III breast cancer or stage I-III ovarian cancer; all antitumor therapies, excluding hormonal therapy, have been completed at least 60 days prior to enrollment
* ECOG Performance Status 0-1 (within 90 days of enrollment)
* Sedentary: <90 minutes/week of moderate-intensity (not exhausting, light perspiration, e.g. fast walking, tennis, easy bicycling, easy swimming, popular and folk dancing) physical activity during the preceding 2 months, and <30 minutes/month of any high-intensity activity (heart beats rapidly, sweating, e.g. running, aerobics classes, cross country skiing, vigorous swimming, vigorous bicycling) in the past 2 months

Exclusion Criteria:

* Evidence of active malignant disease
* Currently has breast implant (which limits the performance of many yoga poses)
* Significant cardiopulmonary disease, severe arthritis, glaucoma or any other medical conditions that make yoga practice unsafe as determined by a study investigator.
* Patient requires regular use of beta blockers or calcium channel blockers.
* Use of any medication that would interfere with the study's initial blood tests, including insulin or insulin secretagogues, corticosteroids, daily use of NSAIDs (except aspirin at no more than 81 mg/day) within 7 days of the initial study blood test.
* Unlikely to be compliant with the study intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
feasibility of a supervised vigorous yoga practice by the number of patients that complete study. | 2 years
  The study will be deemed feasible and safe if at least 15/20 patients in each arm complete the study. If the underlying feasibility rate is 90%, then the probability of 15/20 patients or more completing the study is 98.9%, and 97.8% for 15/20 patients completing in the study in both arms simultaneously.
safety of a supervised vigorous yoga practice by the number of serious adverse events reported. | 2 years
  Each serious adverse event (SAE), defined as grade III or IV toxicity, will be evaluated by the PI or a Co-PI and its relationship to the study intervention is determined by the PI or a Co-PI. The study will be deemed feasible and safe if at least 15/20 patients in each arm complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deng, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Deng G, Bao T, Ryan EL, Benusis L, Hogan P, Li QS, Dries A, Konner J, Ahles TA, Mao JJ. Effects of Vigorous Versus Restorative Yoga Practice on Objective Cognition Functions in Sedentary Breast and Ovarian Cancer Survivors: A Randomized Controlled Pilot Trial. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221089221. doi: 10.1177/15347354221089221. PMID 35861215
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/